CLINICAL TRIAL: NCT05095545
Title: Multi-center, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study to Assess the Efficacy and Safety of the AV5080 Drug in Patients With Influenza
Brief Title: Dose Range Study to Evaluate the Efficacy and Safety of AV5080 in Patients With Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLU-AV5080-02
Record Dates: First submitted 2021-10-22; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Influenza
Keywords: Influenza treatment in adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study was double-blinded. The staff of the clinical sites and the patients were unaware of the treatment and its doses assigned to each specific patient. Blinding was provided by a placebo mask (each patient received capsules containing either 80 mg of AV5080 or placebo), and drug distribution was controlled by the IWRS. Each patient was given two bottles containing the capsules, a bottle A and a bottle B. The two bottles had the same number and differed in lettering and label color: the bottle A had a white label and the bottle B had a yellow label. Patients were to take one capsule in the morning - from bottle A, and one capsule in the evening - from the bottle B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): AV5080 80 mg"/day (80 mg in the morning + placebo in the evening)
  Interventions: Drug: AV5080
- Group 2 (Experimental): AV5080 160 mg"/day (80 mg in the morning + 80 mg in the evening)
  Interventions: Drug: AV5080
- Group 3 (Placebo Comparator): "Placebo" (placebo in the morning + placebo in the evening)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AV5080 — Hard gelatin capsules with a white body
  Arms: Group 1; Group 2
Other: Placebo — Hard gelatin capsules with a white body
  Arms: Group 3

SUMMARY:
Assessment of the effect reached with the different doses of AV5080 on the duration and severity of influenza symptoms based on the incidence of their resolution within 96 hours from study treatment initiation compared to Placebo.

The absence of influenza symptoms or their reduction to mild severity for at least 24 hours indicates the resolution of influenza.

DETAILED DESCRIPTION:
The study was a multi-center, double-blind, randomized, parallel- group clinical study to assess the efficacy and safety of different AV5080 doses as compared to placebo in patients with influenza during the 5-day treatment period.

The study included only patients with influenza of mild and moderate severity, without complications, both outpatients and those hospitalized for epidemiological reasons. The study included three periods for each patient: Screening, randomization, and study treatment, follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. Males and females between 18 and 65 years old (inclusive);
3. Outpatients and those hospitalized for epidemiological reasons with mild and moderate severity diagnosed influenza (ICD 10: J10 Influenza caused by an identified influenza virus) without complications; The severity of influenza is defined under the Influenza in the Influenza in Adults Clinical Guidelines of the National Scientific Society of the Infectious Diseases Specialists;
4. Positive enzyme-linked immunosorbent assay for influenza virus at screening;
5. At least one episode of an increased body temperature up to 38°C and above within 48 hours before screening;
6. The presence of at least one of the following symptoms of moderate severity on screening: Headache, weakness/malaise, myalgia/muscle ache, hot flash/chills;
7. Duration of the disease not exceeding 48 hours (according to the patient) on screening;
8. Consent of patients to use adequate contraception methods throughout the study. Adequate contraception methods include:

   * Oral contraceptives or contraceptive patches;
   * Condoms or diaphragms (barrier method) with spermicide; or
   * An intrauterine device.

Exclusion Criteria:

1. Pregnant or breastfeeding women or women planning to become pregnant during the clinical study; women of child-bearing potential (including women in their post-menopausal period for less than two years) who do not use adequate contraception measures;
2. Individual intolerance of the AV5080 drug or its components;
3. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption;
4. Influenza complications, signs of a bacterial infection or severe disease course at the screening (based on the criteria specified in the Influenza in Adults Clinical Guidelines of the National Scientific Society of Infectious Diseases Specialists, 2014);
5. The history of anti-influenza immunization within 12 months before the screening;
6. Participation in other clinical studies within three months before screening;
7. Chronic respiratory system diseases (asthma, COPD);
8. Administration of neuraminidase inhibitors (zanamivir, oseltamivir), immunomodulators, systemic glucocorticoids, and antibiotics within one month before screening;
9. HIV infection, chronic hepatitis С or hepatitis B infection (according to the patient's history);
10. Significant cardiovascular diseases at present or within 12 months prior to screening including: class III or IV chronic heart failure (as defined by NYHA), severe arrhythmia requiring administration of class Ia, Ib, Ic or III anti-arrhythmic drugs, non-stable angina, myocardial infarction, previous surgery on the heart and coronary vessels, significant heart valves diseases, transient ischemic attack or stroke, uncontrollable hypertension with systolic BP > 180 mmHg and diastolic BP > 110 mmHg, pulmonary embolism or deep vein thrombosis;
11. Chronic alcohol abuse, drug abuse or addiction to the other chemicals in history;
12. Inability to read or write; unwillingness to understand and comply with the Protocol procedures; non-compliance with the drug dosing regimen or procedures which, in the Investigator's opinion, may affect the study results or the patient's safety and prevent the patient to participate in the study; any other concomitant diseases or severe mental disorders, which make the patient ineligible to participate in the study, limit the legal basis for Informed Consent procedure, or may affect the patient's ability to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who reported resolution of influenza symptoms within 96 hours from the start of therapy | 30 days
  The absence of influenza symptoms or their reduction to mild severity for at least 24 hours indicates the resolution of influenza.

SECONDARY OUTCOMES:
Time to symptoms resolution | 30 days
  The time before the resolution of influenza symptoms
Incidence rate of influenza virus elimination until Day 6 | 6 days
  The incidence rate of influenza virus elimination from mucous membranes of the nasopharynx and oropharynx until Day 6
Change in titer of antibodies on Day 15 compared to baseline; | 15 Days
  Change in titer of IgG and IgM antibodies to influenza A and B virus on Day 15 compared to baseline;
The incidence rate of influenza complications | 29 Days

CONTACTS AND LOCATIONS:
Locations (10):
- Russia (10):
  - City polyclinic №10, Kazan'
  - Infectious Clinical Hospital No. 1 of the Moscow City Health Department, Moscow
  - GBUZ NO Infections Clinical Hospital No.2, Nizhny Novgorod
  - Podolsk City Clinical Hospital №3, Podolsk
  - City Hospital No. 1 n.a. ON. Semashko, Rostov-on-Don
  - City Clinical Hospital of Infectious Diseases No. 17, Saint Petersburg
  - City hospital №40, Saint Petersburg
  - Federal Research Center Institute of Cytology and Genetics, Siberian Branch of the Russian Academy of Sciences, Stavropol
  - Voronezh Regional Clinical Infectious Diseases Hospital, Voronezh
  - Medical Center for Diagnostics and Prevention Plus, LLC, Yaroslavl

IPD SHARING:
Plan to Share IPD: No